CLINICAL TRIAL: NCT03896919
Title: Impact of HLA-DQ Mismatch on Acute Rejection of Kidney Transplantation
Brief Title: HLA-DQ in Acute Kidney Transplantation Rejection
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maha Gamal Ahmed, principle investigator, Assiut University
Other Study IDs: HLA-DQ in kidney transplant.
Record Dates: First submitted 2019-03-26; First posted 2019-04-01 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases: HLA-DQ mismatched recipient-donor pairs
  Interventions: Diagnostic Test: HLA-DQ by luminex technology in kidney transplantation
- control: HLA-DQ matched recipient- donor pairs
  Interventions: Diagnostic Test: HLA-DQ by luminex technology in kidney transplantation

INTERVENTIONS:
Diagnostic Test: HLA-DQ by luminex technology in kidney transplantation — HLA typing (DQ) for donor and recipient using Luminex microbead method from EDTA blood sample

SUMMARY:
- Study the impact of HLA-DQ mismatch on acute rejection of Kidney transplantation

DETAILED DESCRIPTION:
Introduction Human Leukocyte Antigens (HLA). The major histocompatibility complex (MHC) is a gene region coding for cell surface proteins important for the immune system. MHC is the most complex immunogenetic system presently known in humans . HLA are groups of cell surface proteins encoded by genes in MHC which are known as HLA in humans and H-2 in mice .

HLA genes are located on the short arm of chromosome 6 at 6p21 position , occupying a genetic region of 4Mbps. The human immune system uses HLA's uniqueness to distinguish self from non-self. HLA are responsible for the presentation of "foreign" peptides (antigens) to the immune competent cells. T lymphocytes recognize foreign antigens only when it combines with HLA molecules.

Humans have three class I HLA (A, B, C) that are present on all nucleated cells and six class II HLA (DPA1, DPB1, DQA1, DQB1, DRA, DRB1) that are present only on antigen-presenting cells and lymphocytes. Three of the seven heterodimers (HLA-A, -B, and -DRB1) contribute to the majority of immunogenicity of mismatched antigens and therefore traditional HLA-typing methods have primarily focused on these alleles .

Renal transplantation is the gold standard therapeutic strategy of replacing renal dysfunctions that offers the best survival to the patients with end-stage renal disease (ESRD). Kidney transplantation is associated with 68% lower risk of death than dialysis . Graft and patient survival after kidney transplantation have improved over the past decade. Death-censored graft survival has increased steadily over the past decade in both adults and pediatric recipients. Data provided by the Scientific Registry of Transplant Recipients (SRTR) demonstrate a 10-year overall graft survival for both living and deceased donors of approximately 55 to 60 percent compared with 35 to 40 percent from a decade prior .

Renal transplantation success is dependent on the reaction of the immune system primarily against human leucocyte antigen (HLA) proteins of the transplant. Patients previously exposed to non-self HLA through transplant, blood transfusions or pregnancy may develop antibodies reactive to HLA .

HLA matching provides beneﬁts in improving outcomes in kidney transplantation and remains part of the kidney allocation. HLA-DR matching has a much greater effect on graft outcomes compared with matching at the HLA-A or -B locus.

Although HLA-DQ does not factor into organ allocation, its relative importance has been increasingly recognized. Recipients with de novo anti-DQ donor-speciﬁc antibodies have a higher incidence of acute rejection, transplant glomerulopathy, and graft loss . The effect of broad antigen HLA-DQ mismatching on kidney transplantation has not been clearly established. Although older studies found no signiﬁcant correlation between HLA-DQ mismatching and graft outcomes , more recent data from the Australia and New Zealand Dialysis and Transplant Registry suggested that HLA-DQ mismatching affects outcomes .

Broad antigen HLA-DQ matching between each recipient and donor on the basis of serologic typing is available for the majority of kidney transplant recipients in the United Network for Organ Sharing (UNOS) registry . Using UNOS data, the investigators sought to determine the effect of HLA-DQ matching on acute rejection and graft loss after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* The patients who will receive renal transplants.

Exclusion Criteria:

* Recipients with pre-transplantation desensitization protocols.
* Recipients with history of previous transplant or pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will be carried out on (30) renal transplant Recipient- Donor pairs who will be recruited from transplantation unit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Combined incidence of DSA or IA on peripheral blood molecular profiling | Baseline
  DSA considered as a binary variable (positive or negative), with positivity based on a threshold criteria of Mean Fluorescence Intensity (MFI) approaching 1000. IA will be considered present or absent using a molecular assay.

SECONDARY OUTCOMES:
Incidence of HLA-DQ DSA [ Time Frame: assessed at days 3,7,15,30 post transplantation | baseline
  Human Leukocyte Antigen, Class II, DQ locus DSA (HLA-DQ DSA). Assessed in subjects who are DSA positive

CONTACTS AND LOCATIONS:
Overall Officials: sohair k sayed, prof.doctor, Study Director — clinical pathology
Locations (1):
- Assiut U, Asyut, Egypt

REFERENCES:
- See also: Clinical issues in renal transplantation in the elderly. Clin Transplant 2015; 29: 167-175 — https://www.ncbi.nlm.nih.gov/pubmed?cmd=search&term=HOD+T%5Bau%5D&dispmax=50
- See also: The association between broad antigen HLA mismatches, eplet HLA mismatches and acute rejection after kidney transplantation. Transplant Direct 2: e120, 20 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5862565/
- See also: donor-speciﬁc HLA-DQ antibodies may contribute to poor graft outcome after renal transplantation. Kidney Int 82: 598-604, 2012 . — https://www.ncbi.nlm.nih.gov/pubmed/22622504